CLINICAL TRIAL: NCT00171587
Title: A Phase IB, Open-label, Dose-escalating Study of Vatalanib in Combination With Capecitabine in Patients With Advanced Cancer
Brief Title: Study of the Safety, Tolerability, Pharmacokinetics, and Anti-tumor Effects of Vatalanib in Combination With Capecitabine in Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Bayer (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPTK787 0134/306220
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2009-11-19 (Estimated); Status verified 2009-11

CONDITIONS: Tumors; Neoplasm Metastasis
Keywords: Metastatic solid tumors; PTK787/ZK 222584; Vatalanib; Capecitabine; VEGF (vascular endothelial growth factor); Histologically confirmed metastatic solid tumors
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis | interventions — vatalanib

INTERVENTIONS:
Drug: PTK787/ZK 222584 (vatalanib)

SUMMARY:
The objective of this study is to assess the safety, tolerability, dose limiting toxicity, and maximum tolerated dose of vatalanib administered orally once daily in combination with capecitabine in patients with advanced cancer. The study is also designed to determine the effect of vatalanib on the pharmacokinetics of capecitabine and the effect of capecitabine on the pharmacokinetics of vatalanib, and to describe the anti-tumor activity of this combination regimen.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed advanced cancer that is refractory to standard therapy or for which no standard therapy exists (for dose escalation phase of the study only)
* Patients with histologically confirmed metastatic solid tumors or colorectal cancer presenting with metastatic disease and who received up to four prior chemotherapies for metastatic disease (for dose expansion phase of the study only)
* Measurable or non-measurable disease as determined by Response Evaluation Criteria in Solid Tumors (RECIST) criteria
* Age >= 18 years old
* Karnofsky Performance Status (KPS) of >= 70
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L
* Hemoglobin (Hgb) >= 9 g/dl
* Platelets >= 100 x 10^9/L
* Aspartate aminotransferase (AST/SGOT) and alanine aminotransferase (ALT/SGPT) <= 3.0 x upper limit of normal (ULN)
* Serum bilirubin <= 1.5 x ULN
* Serum creatinine <= 1.5 x ULN and 24-hour creatinine clearance >= 50 ml/min
* Total urinary protein in a 24-hour urine collection <= 500 mg
* Life expectancy of greater than 3 months
* Written informed consent obtained according to local guidelines

Exclusion Criteria:

* Patients who have acute or chronic leukemias, lymphoma, or multiple myeloma
* Patients who have known bone marrow involvement with tumor
* Patients with a history of primary central nervous system tumors or brain metastases
* Prior allogeneic, syngeneic, or autologous bone marrow transplant or stem cell transplant
* Patients who have had more than two prior chemotherapy regimens for metastatic disease (for dose escalation phase of the study only)
* Patients who have received chemotherapy less than 4 weeks (6 weeks for nitrosoureas or mitomycin-C and 2 weeks for vincristine) prior to entry on this study or who have not recovered from side effects of such therapy
* Patients who have received immunotherapy within 2 weeks or who have not recovered from side effects of such therapy
* Patients who have received radiotherapy within 2 weeks or who have not recovered from side effects of such therapy. The site of radiotherapy should not be the only site of measurable disease.
* Major surgery within 2 weeks prior to entry on this study or patients who have not recovered from side effects of such therapy
* Patients who have received investigational drugs within 4 weeks prior to entry on this study or who have not recovered from side effects of such therapy
* Patients who are pregnant or breast feeding, or adults of reproductive potential not employing an effective method of birth control. Oral, implantable, or injectable contraceptives are not considered an effective method of birth control for this study. (Women of childbearing potential must have a negative serum pregnancy test 48 hours prior to administration of chemotherapy).
* Concurrent severe and/or uncontrolled medical disease (i.e., uncontrolled diabetes, congestive cardiac failure, myocardial infarction within 6 months, poorly controlled hypertension, history of labile hypertension, history of poor compliance with antihypertensive regimen, chronic renal disease, or active uncontrolled infection) which could compromise participation in the study
* Acute or chronic liver disease (e.g., hepatitis, cirrhosis)
* Confirmed diagnosis of HIV infection
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of PTK787/ZK 222584 (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, bowel obstruction, or inability to swallow the capsules/tablets)
* Patients who are taking Coumadin (warfarin sodium)
* Patients unwilling to or unable to comply with the protocol

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2002-05; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Safety
Tolerability

SECONDARY OUTCOMES:
Pharmacokinetics

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Chair — Novartis
Locations (1):
- University of Chicago, Chicago, Illinois, United States